CLINICAL TRIAL: NCT05719753
Title: A Pilot Study to Characterise the Effectiveness of a Bacteriophobic Coating in Preventing
Brief Title: The Effectiveness of a Bacteriophobic Coating on Urinary Catheters
Acronym: PRO033CSP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Camstent Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 18057
Record Dates: First submitted 2022-12-27; First posted 2023-02-09 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2020-08

CONDITIONS: Urinary Tract Infections
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Placebo Comparator): Bard Catheter
  Interventions: Device: Standard Care
- Camstent Coated Catheter (Experimental): The Camstent Coated Foley Catheter is an all-silicone two-way Foley-type urinary catheter, to which a proprietary polymeric coating has been applied.
  Interventions: Device: Camstent Coated Catheter

INTERVENTIONS:
Device: Camstent Coated Catheter — The Camstent Coated Foley Catheter is an all-silicone two-way Foley-type urinary catheter, to which a proprietary polymeric coating has been applied.
  Arms: Camstent Coated Catheter
Device: Standard Care — Bard Catheter
  Arms: Standard of Care

SUMMARY:
To assess if a bacteriophobic coating prevents biofilm and host protein accumulation on urinary catheters and inflammatory protein release in urine following catheterization

DETAILED DESCRIPTION:
The purpose of the study is to provide pilot information on the characteristics of the biofilm formed on the coated catheter compared to a standard catheter. The two objectives are;

1. to evaluate the catheter's on-label performance in customary clinical use.
2. to quantify biofilm formation on the catheter surface, and to compare it with biofilm formation on the hospitals current uncoated catheters.

ELIGIBILITY:
Inclusion Criteria:

1. All patients undergoing colorectal resection routinely requiring a urinary catheter as part of their standard post-operative care.
2. Patients aged 18-85 years will be eligible for the study.
3. Able to give informed consent.

Exclusion Criteria:

1. Patients that have or recently (within 3 weeks) had a urinary catheter, or those with signs of current urinary tract infection.
2. Pregnant patients.
3. Patients with a potentially immunocompromised condition (steroids, HIV)
4. Patients who are unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2021-09-20 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
An analytic characterisation of catheters after routine patient use, will yield estimates of the difference in biofilm density between coated and non-coated catheters. | 1 year
  An analytic characterisation of catheters after routine patient use, will yield estimates of the difference in biofilm density between coated and non-coated catheters.

SECONDARY OUTCOMES:
catheter blockage | 1 year
  catheter blockage
catheter associated infection | 1 year
  catheter associated infection
Ease of insertion and removal of the catheter since it creates a very smooth and slippery surface using the NHS staff standard clinical feedback form. | 1 year
  Ease of insertion and removal of the catheter since it creates a very smooth and slippery surface using the NHS staff standard clinical feedback form.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Nottingham, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided